CLINICAL TRIAL: NCT01829919
Title: Evaluation of Pharmacokinetics of Paroxetine Following Single and Repeat Oral Administration of Mesafem (7.5 mg Paroxetine Mesylate) Capsules in Healthy Postmenopausal Women
Brief Title: Pharmacokinetic Evaluation of Brisdelle™ (Formerly Known as Mesafem) Following Single & Repeat Oral Administration in Healthy Postmenopausal Women
Acronym: N30-005
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N30-005
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Postmenopausal Symptoms
Keywords: Menopause; Hot flashes; Vasomotor symptoms; Climacteric symptoms; perimenopause; Mesafem; Brisdelle; Low-Dose Mesylate salt of Paroxetine (LDMP)
MeSH Terms: conditions — Hot Flashes | interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brisdelle (paroxetine mesylate) (Experimental): Brisdelle (paroxetine mesylate) Capsules taken orally with 240 mL of water for 20 days.
  Interventions: Drug: Brisdelle (paroxetine mesylate)

INTERVENTIONS:
Drug: Brisdelle (paroxetine mesylate) — All subjects will receive Brisdelle (paroxetine mesylate) Capsules 7.5 mg, first as a single dose and then, following a five-day wash-out period, once per day for 14 days.
  Other Names: Former Names: Mesafem capsules 7.5 mg or; LDMP (Low-Dose Mesylate salt of Paroxetine)

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (absorption, breakdown and elimination from the body), safety and tolerability of Brisdelle (paroxetine mesylate) Capsules 7.5 mg when given as a single dose and multiple doses.

DETAILED DESCRIPTION:
This study is for research only and is not designed to treat a medical condition.

ELIGIBILITY:
Inclusion Criteria:

Subjects who are healthy postmenopausal, non-smoking women of any race and ≥40 years of age at screening.

Exclusion Criteria:

Subjects who have a recent history or presence of glaucoma, migraines, cardiovascular, hepato-biliary, renal, gastrointestinal, neurologic, psychiatric, dermatologic, pulmonary, cerebrovascular, endocrine, hematologic, thromboembolic, immunologic disease or any other disorder which requires physician care; subjects who have existing medical conditions which might interfere with absorption, distribution, metabolism, or excretion of study medication; history of self-injurious behavior; history of clinical diagnosis of depression; or treatment for depression; history of clinical diagnosis of border-line personality disorder; presence of any of the following psychiatric disorders within the timeframes specified: Major Depressive Disorder-Lifetime; Dysthymia-Past 2 Years; Bipolar Disorder-Lifetime; Panic Disorder-Lifetime; Agoraphobia-Past Month; Social Phobia-Past Month; Obsessive Compulsive Disorder-Past Month; Generalized Anxiety-Lifetime; Psychotic Disorders-Lifetime; Anorexia Nervosa-Past 10 Years; Bulimia-Past 10 Years; Suicidality/Suicide Ideation-Lifetime; Post Traumatic Stress Disorder-Lifetime.

Subjects with a history of seizures; sitting blood pressure (BP) < 90/50 or > 150/90 mmHg; sitting heart rate (HR) < 45 or > 90 beats/min; clinical laboratory test results outside of the normal range for the laboratory conducting the test; positive urine pregnancy test at Screening or Day 0; subjects who have a history of sensitivity to active and/or inactive ingredients in Brisdelle (paroxetine mesylate) Capsules 7.5 mg; subjects who have a history of significant allergies; subjects who have a present or past history of narcotic addiction, drug abuse, or alcoholism; subjects who have smoked or used tobacco during the last 6 months; subjects who have donated one or more pints of blood within 30 days prior to treatment administration; subjects who have symptoms of any significant acute illnesses at the screening visit; subjects who used any investigational drug within 30 days prior to treatment administration; subjects who took any substances known to be Cytochrome P450 2D6 (CYP2D6) inhibitors within 14 days of study start and throughout the entire study; subjects who used any prescription medications within 14 days of the screening visit; subjects who used St John's Wort within 14 days of the screening visit; subjects who used any over the counter preparations including herbal or nutritional supplements and multivitamins within 10 days prior to receiving the first study treatment; subjects who have consumed foods or beverages containing caffeine/xanthine or alcohol; subjects who have a positive screen for hepatitis B surface antigen (HBsAg) or hepatitis C antibody; subjects who have a positive screen for the Human Immunodeficiency Virus (HIV) antibody; subjects who have a positive urine drug screen; subjects who have any clinically significant illness within 90 days prior to receiving the first dose of study medication.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, MD, Principal Investigator
Locations (1):
- SNBL Clinical Pharmacology Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Cristina Castelli M, Bhaskar S, Lippman J. Pharmacokinetic properties of once-daily oral low-dose mesylate salt of paroxetine (LDMP 7.5 mg) following single and multiple doses in healthy postmenopausal women. Clin Ther. 2013 Jun;35(6):862-9. doi: 10.1016/j.clinthera.2013.05.001. PMID 23795577
- See also: Sponsor — http://www.noven.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg: Brisdelle (paroxetine mesylate) Capsules 7.5 mg
  All subjects will receive Brisdelle (paroxetine mesylate) Capsules 7.5 mg, first as a single dose and then, following a five-day wash-out period, once per day for 14 days.
Period: Overall Study
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 24
Groups:
- Brisdelle (Paroxetine Mesylate) Capsules: Brisdelle (paroxetine mesylate) Capsules
  All subjects will receive Brisdelle (paroxetine mesylate) capsules, first as a single dose and then, following a five-day wash-out period, once per day for 14 days.
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (7.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: AUC (Hour*ng/mL) Single Dose Pharmacokinetics of Brisdelle™ (Paroxetine Mesylate) Capsules 7.5 mg
Time Frame: Day 1
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Mean (Standard Deviation); unit: Hour*ng/mL
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
Hour*ng/mL
  AUC0-last (Hour x ng/mL) | 86.95 (166.19)
  AUC0-inf (Hour x ng/mL) | 78.80 (189.88)
  AUC0-24 (Hour x ng/mL) | 38.90 (51.83)

2. Primary Outcome: Cmax (ng/mL) Single Dose Pharmacokinetics of Brisdelle™ (Paroxetine Mesylate) Capsules 7.5 mg
Time Frame: Day 1
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
ng/mL | 2.77 (3.38)

3. Primary Outcome: Kel (Hour^-1) Single Dose Pharmacokinetics of Brisdelle™ (Paroxetine Mesylate) Capsules 7.5 mg
Time Frame: Day 1
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Mean (Standard Deviation); unit: Hour^(-1)
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
Hour^(-1) | 0.05 (0.01)

4. Primary Outcome: Mean t1/2 Single Dose Pharmacokinetics of Brisdelle™ (Paroxetine Mesylate) Capsules 7.5 mg
Time Frame: Day 1
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
Hours | 17.30 (11.45)

5. Primary Outcome: Median t1/2 Single Dose Pharmacokinetics of Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Time Frame: Day 1
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Median (Full Range); unit: hours
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
hours | 6.00 [1.00 to 8.00]

6. Primary Outcome: AUC (Hour*ng/mL) Multiple Dose Pharmacokinetics of Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Time Frame: Day 19
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Mean (Standard Deviation); unit: Hour*ng/mL
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
Hour*ng/mL
  AUC0-last (Hour x ng/mL) | 237.34 (222.65)
  AUC0-24 (Hour x ng/mL) | 237.28 (222.64)

7. Primary Outcome: Cmax (ng/mL) Multiple Dose Pharmacokinetics of Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Time Frame: Day 19
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
ng/mL | 13.10 (11.92)

8. Primary Outcome: Cmin (ng/mL) Multiple Dose Pharmacokinetics of Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Time Frame: Day 19
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
ng/mL | 7.67 (7.57)

9. Primary Outcome: Tmax (Hour) Multiple Dose Pharmacokinetics of Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Time Frame: Day 19
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Mean (Full Range); unit: Hours
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
Hours | 6.00 [3.00 to 8.00]

10. Primary Outcome: Accumulation Index Multiple Dose Pharmacokinetics of Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg at Day 19
Description: Accumulation Index is the ratio of AUC 0-24 after multiple doses versus a single dose. It is the increase in drug plasma concentration after multiple dosing until a steady state is reached. In this case the steady state Accumulation Index was calculated at Day 19. Accumulation Index is calculated at the end of the dosing period.
Time Frame: Day 19
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Mean (Full Range); unit: Ratio
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
Ratio | 9.71 [0.12 to 23.48]

11. Primary Outcome: Fluctuation Index (%) Multiple Dose Pharmacokinetics of Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Description: Fluctuation Index is (Cmax-Cmin)/Cavg,ss. It is peak trough fluctuation within one dosing interval at steady state.
Time Frame: Day 19
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Mean (Full Range); unit: Percentage of steady state concentration
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
Percentage of steady state concentration | 75.76 [35.57 to 153.20]

12. Primary Outcome: Cavg,ss (ng/mL) Multiple Dose Pharmacokinetics of Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Time Frame: Day 19
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
ng/mL | 9.89 (9.28)

13. Primary Outcome: Ct (ng/mL) Multiple Dose Pharmacokinetics of Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Description: C(t) is the measured plasma level "Concentration" of the drug at "time = t" expressed as nanograms per milliliter.
Time Frame: Day 19
Population: Safety and evaluable pharmacokinetic populations = 24 randomized subjects.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules 7.5 mg
Number analyzed (Participants) | 24
ng/mL
  Cτ18 (ng/mL) | 8.53 (9.17)
  Cτ19 (ng/mL) | 8.35 (8.49)
  Cτ20 (ng/mL) | 8.79 (9.19)

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 23/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brisdelle (Paroxetine Mesylate) Capsules (N=24)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (7)
Abnormal dreams (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other